CLINICAL TRIAL: NCT04385472
Title: Musculoskeletal Imaging of Runners
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Professor Alister Hart, Professor of Orthopaedics, Royal National Orthopaedic Hospital NHS Trust
Other Study IDs: 13823/001
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Musculoskeletal Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: 3T MRI — The main method used will be 3 Tesla MRI, which is a high resolution imaging technique. The participants will be asked to undergo musculoskeletal MRI scanning (pelvis and lumbar spine).MRI is a non-invasive procedure which excludes the risk of radiation (in comparison to other imaging modalities: X-ray, CT

SUMMARY:
The investigators aimed to assess the impact of long-distance running on musculoskeletal system of runners, by doing high resolution magnetic resonance imaging analysis before and after marathon running.

DETAILED DESCRIPTION:
Rationale for the study: This research will examine a key modifiable risk factor for health and well- being: exercise. Regular exercise is highly recommended by healthcare professionals because the whole body benefits, including cardiorespiratory, musculoskeletal systems and mental wellbeing. Long-distance running is a popular physical activity with more than 30 million individuals running marathons each year. The increasing participation of first-time runners, including older people, has been linked to a rise in related injuries. The ideal dose of exercise is not known and overdosage affects some musculoskeletal tissues and joints more than others. Overdoing a specific amount of exercise and the presence of chronic injuries may pose a great risk on the joints, leading to serious conditions such as osteoarthritis, musculoskeletal injuries, tendinopathy. However, it is not yet clear whether a high dose of exercise such as marathon running damages the musculoskeletal system and there is a growing need for research in the area of running science to better understand this.

Aim: This research aims to do musculoskeletal imaging before and after long-distance running using 3 Tesla magnetic resonance imaging and to provide evidence on how much exercise people should undertake and how to minimise injury.

ELIGIBILITY:
Inclusion Criteria:

* no previous marathon participations
* no present or previous history of hip injuries or surgeries
* asymptomatic hip joints
* no contradindications to hip MRI scanning

Exclusion Criteria:

* pregnant or breastfeeding women
* individuals aged <18 years
* claustrophobia
* history of anxiety or panic attacks
* known hip problems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: asymptomatic long-distance runners
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in radiographic score after marathon running | up to 1 year
Change in self-reported hip questionnaire after marathon running | up to 1 year

SECONDARY OUTCOMES:
Number of participants who finished the training for/and the marathon vs not finishing | up to 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal National Orthopaedic Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided